CLINICAL TRIAL: NCT02249455
Title: Effectiveness of Acapella and ELTGOL (Expiration in Lateral Position With Open Glottis)Technique to Promote Airway Clearance in COPD Patients:a Comparative Study
Brief Title: Effectiveness of Acapella and ELTGOL Technique to Promote Airway Clearance in COPD:a Comparative Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: PSG College of Physiotherapy (Other)
Responsible Party: Principal Investigator, STEFFI VARGHESE P, post graduate in cardiopulmonary rehabiltation, PSG College of Physiotherapy
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 14\305
Record Dates: First submitted 2014-09-04; First posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Exhalation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Acapella (Experimental): Acapella is given to the patients twice daily for 20 min.
  Interventions: Device: Acapella
- ELTGOL (Experimental): Expiration with open glottis in lateral position is done twice daily for 20 min
  Interventions: Other: ELTGOL
- conventional physiotherapy (Active Comparator): Conventional physiotherapy like breathing exercise, active coughing, chest mobilisation was encouraged twice daily for 20 min.
  Interventions: Other: conventional physiotherapy

INTERVENTIONS:
Device: Acapella — Treatment time for 20 min twice daily
  Other Names: ACAPELLA DHD
  Arms: Acapella
Other: ELTGOL — ELTGOL technique 20 min twice daily
  Other Names: Expiration in lateral position with open glottis for twenty min twice daily.
  Arms: ELTGOL
Other: conventional physiotherapy — Conventional physiotherapy was given twice daily for 20 min
  Arms: conventional physiotherapy

SUMMARY:
To compare the efficacy of acapella and expiration against open glottis (ELTGOL) technique in promoting airway clearance of chronic obstructive pulmonary disease (COPD) patients

DETAILED DESCRIPTION:
This study is carried out to determine the effectiveness of acapella and expiration in lateral position with open glottis to clear the secretion in COPD patients. The sessions will be carried twice daily for twenty minutes. The outcome measures are values of pre and post intervention fev1/fvc and breathlessness cough sputum scale. Duration of the study will be for five days.

ELIGIBILITY:
Inclusion Criteria:

* Mild copd
* Moderate copd
* Patient able to sustain expiratory flow greater than 15l/min
* Patient expectorate more than 25.-30ml

Exclusion Criteria:

* Severe copd
* Peripheral oxygen saturation lower than 85%
* Rr>35breaths/min
* Current acute chest pain
* Recent history of haemoptysis

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-07; Primary Completion 2014-12 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Change in Force expiratory volume in one second | change from baseline at 30 minutes
  Fev1/fvc values were noted after pre and post intervention of airway clearance manoeuver

SECONDARY OUTCOMES:
Change in breathlessness cough sputum score | change from baseline at 5 days
  Bcss scale was interviewed to the patient on first day and the fifth day. The changes were noted.

CONTACTS AND LOCATIONS:
Overall Officials: steffi varghese, mpt, Principal Investigator — psg ims&r
Locations (1):
- Steffi Varghese, Coimbatore, Tamil Nadu, India